CLINICAL TRIAL: NCT06598956
Title: An Open, Parallel, Single-dose Phase I Clinical Study to Evaluate the Pharmacokinetics and Safety of TQ05105 Tablets in Patients With Different Levels of Renal Function
Brief Title: To Evaluate the Pharmacokinetics and Safety of TQ05105 Tablet in Renal Impairment Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-I-06
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-09

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild Renal Impairment(GFR:60~89 mL/min) (Active Comparator): 15 mg orally , single dose
  Interventions: Drug: TQ05105
- Moderate Renal Impairment(GFR:30~59 mL/min) (Active Comparator): 10 mg orally , single dose
  Interventions: Drug: TQ05105
- Severe Renal Impairment(GFR:15~29 mL/min) (Active Comparator): 5 mg orally , single dose
  Interventions: Drug: TQ05105
- Normal(GFR≥90mL/min) (Active Comparator): 15 mg orally , single dose
  Interventions: Drug: TQ05105

INTERVENTIONS:
Drug: TQ05105 — TQ05105 is a Janus kinase (JAK) and Rho-associated coiled-coil-containing protein kinase (ROCK) inhibitors.

SUMMARY:
This is an open, open-label, parallel, single-dose, phase I clinical study designed to evaluate the pharmacokinetic (PK) profile of TQ05105 tablet in patients with renal impairment after a single dose, and to evaluate the urinary excretion of the drug in these patients after a single dose, as well as to evaluate the safety of the drug in these patients after a single dose.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet all of the following criteria for inclusion in this study:

* Understand the content, process and possible adverse reactions of the trial, be able to complete the study in accordance with the requirements of the trial protocol, and voluntarily sign the informed consent;
* Participants (including their partners) voluntarily used effective contraception within 6 months from screening until the last use of study drug;
* Participants aged 18 ~ 75 ;
* Body mass index (BMI) and 18 or 32 kg/m2 or less, and the male weight 50 kg or greater, female weight 45 kg or more;

For renal impairment subjects, also required meet all of the following criteria for inclusion in this study:

* Subjects with moderate to severe renal insufficiency and end-stage renal disease were required to meet the diagnostic criteria for chronic kidney disease;
* Stable renal function: creatinine detection of at least two intervals of 3 days (30 days before the screening test results for the first time acceptable) inside and outside school or in our test result, and two detecting serum creatinine results before and after the fluctuation (calculation formula: (second results - 1)) / 1 time is less than 30%;
* During the screening period, the individual glomerular filtration rate (GFR, mL/min, using the modification of diet in renal disease (MDRD) formula, based on the results of the second serum creatinine test) was classified as follows: 60≤GFR≤89 mL/min (Group A, mild renal dysfunction, Chronic kidney disease (CKD) 2 period), or 30≤GFR≤59 mL/min (Group B, moderate renal dysfunction, CKD 3 period), or 15≤GFR≤29 mL/min (Group C, severe renal dysfunction, CKD 4 period).

For normal subjects, also required meet all of the following criteria for inclusion in this study:

* During the screening period, normal vital signs, laboratory tests, physical examination, 12-lead ECG, chest radiographs, and echocardiography results, or abnormal results determined by the investigator to be of no clinical significance, are considered normal.
* Individual glomerular filtration rate (GFR, mL/min, using MDRD formula) during the subject screening period: GFR≥90 mL/min.

Exclusion Criteria:

All subjects were not eligible for the study if they met any of the following criteria:

* Individuals with an allergy disposition, or those with a history of allergic reactions to polymyxin-type drugs (including polymyxin B, polymyxin sulfate, and polymyxin E monosodium salt);
* Participants who have had any type of treatment or untreated malignant tumor (excluding basal cell carcinoma of the skin) within the past 5 years or at baseline;
* Participants who have had a serious digestive, respiratory, nervous, hematological, endocrine, tumor, immune, psychological, or cardiovascular disease within the past year and are deemed unfit for the study by the investigator;
* Participants who have had a major illness or surgery within the past 4 weeks or plan to undergo surgery during the study period;
* Participants who have donated blood (or lost blood) of at least 400 mL within the past 3 months or have received blood products;
* Participants who have smoked an average of more than 10 cigarettes per day within the past 3 months;
* Participants who have consumed an average of more than 14 units (female subjects) or 21 units (male subjects) of alcohol per week within the past 3 months (1 unit = 285 mL of beer, 25 mL of distilled spirits, or 100 mL of wine);
* Participants who have consumed a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive tea, coffee, grapefruit/grapefruit juice, and/or caffeine-containing beverages (an average of 8 cups or more per day, 200 mL per cup) within the past 2 weeks;
* Participants who have consumed any alcoholic beverages within 48 hours of receiving the study drug or who have a positive breath alcohol test;
* Individuals with a history of drug abuse within the past 5 years, or who have used soft drugs (e.g. marijuana) within the past 3 months, or who have used hard drugs within the past year, or who have a positive drug screen at baseline;
* Individuals with positive HIV antibody; positive Hepatitis C virus (HCV) antibody or HBsAg positive; positive syphilis treponemal antibody;
* Pregnant or lactating women, and women of childbearing potential with a positive pregnancy test result;
* Individuals who have used strong inhibitors or inducers of liver metabolizing enzymes within the past 14 days;
* Other situations that the investigator considers inappropriate for enrollment.

Renal impairment subjects were not eligible for the study if they met any of the following criteria:

* With acute renal failure, has a history of renal transplantation, or expected during the test need a kidney transplant or accept any type of dialysis patients;
* With obstructive urinary tract diseases (such as urinary tract obstruction caused by urinary calculi, abdominal space occupying lesions, etc.) or causes of renal damage unrelated to renal parenchymal dysfunction (such as polycystic kidney disease, renal tumor, renal artery stenosis, drugs, severe infection, hypovolemia, heart failure, etc.);
* Patients with urinary incontinence;
* Screening, treatment and/or other drug combined treatment of diseases have not meet a month stability, within a month or a new medication (except for temporary or intermittent use of drugs, such as a month use erythropoietin, or temporary require the use of diuretics, etc.);
* Congestive heart failure of New York Heart Association (NYHA) class III or IV, or left ventricular ejection fraction <50% at screening;
* On the stage screening or baseline, systolic blood pressure 160 mmHg and 80 mmHg or less, or diastolic blood pressure 100 mmHg or 50 mmHg or less, or heart rate < 50 times/min or > 100 times/min;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2×Up Limit of Normal(ULN), total bilirubin >1.5×ULN; Albumin < 25 g/L; Absolute neutrophil count <1.0×109/L; Hemoglobin < 80 g/L; The platelet count < 75 x 109 / L;
* Participants who were enrolled in another clinical trial and used any investigational drug or medical device within 3 month before screening, based on the last investigational drug administration date (at least 5 half-lives between investigational drug administration and this study administration for long-half-life investigational drug);

Normal subjects were excluded from the study if they met any of the following criteria:

* Participants who were enrolled in other clinical trials and used any investigational drug or device within 3 months before screening, based on the date of last investigational drug administration (for investigational drug with long half-life, at least 5 half-life intervals between investigational drug administration and this study);
* For 14 days before or within 5 half-life of longer (to) the use of any drugs.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Maximum plasma drug concentration of TQ05105 and TQ12550
Area under the concentration-time curve (AUC) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Area under the plasma concentration-time curve of TQ05105 and TQ12550
Time-to-maximum concentration( Tmax) of TQ05105 and TQ12550 | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Time-to-maximum concentration
Plasma half life (t1/2) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  The time it takes for the concentration or amount in the body of that drug to be reduced by exactly one-half of TQ05105 and TQ12550
Total body clearance (CLt) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Total body clearance of TQ05105 and TQ12550
Renal clearance (CLr) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Renal clearance of TQ05105 and TQ12550
Apparent volume of distribution (Vd/F) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  Volume of distribution based on the terminal phase of TQ05105 and TQ12550
Terminal elimination rate (λz) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  First-order rate constant associated with the terminal (log-linear) elimination phase of TQ05105 and TQ12550
Mean residence time (MRT) | Before administration, 10, 20, 30, 45 minuets，1, 2, 3, 4, 6, 8, 12, 24 hours after administration
  The average time that the drug stays in the body of TQ05105 and TQ12550

SECONDARY OUTCOMES:
Amount Excreted in Urine as Unchanged Drug or Metabolite (Ae0-24) | Before administration, 0~ 3, 3~6， 6~9, 9~12, 12~16, 16~24, 24~36, 36~48 hours after administration
  Ae0-24 of of TQ05105 and TQ12550
Adverse event rate | Baseline up to 72 hours
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital), Jinan, Shandong, China